CLINICAL TRIAL: NCT01988103
Title: A Phase 2B, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) In Japanese Subjects With Moderate-To-Severe Plaque-Type Psoriasis
Brief Title: Efficacy and Safety Study of Two Doses of Apremilast (CC-10004) In Japanese Patients With Moderate-To-Severe Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-011
Record Dates: First submitted 2013-05-24; First posted 2013-11-20 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis; Psoriatic Arthritis; Psoriasis Arthropatica
Keywords: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 20mg (Experimental): Apremilast 20 mg tablets orally twice a day (BID)
  Interventions: Drug: Apremilast; Drug: Placebo
- Apremilast 30mg (Experimental): Apremilast 30 mg tablets orally BID
  Interventions: Drug: Apremilast; Drug: Placebo
- Placebo (Placebo Comparator): Identically-appearing placebo tablets BID for 16 weeks followed by participants being re-randomized in a blinded fasion to apremilast 20 mg or 30mg tablets BID for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — 20 mg tablet BID for 68 weeks
  Other Names: CC-10004; Otzela
  Arms: Apremilast 20mg
Drug: Apremilast — 20 mg tablet BID for 68 weeks
  Other Names: CC-10004; Otzela
  Arms: Apremilast 30mg
Drug: Placebo — Placebo tablet BID for 16 weeks

SUMMARY:
This study will test the clinical effectiveness and safety of two orally administered doses of apremilast compared to placebo in Japanese patients with moderate-to-severe plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a phase 2b, multicenter, randomized, double-blind, placebo-controlled study of the efficacy and safety of apremilast 20 mg twice a day (BID), apremilast 30 mg BID, and placebo in Japanese participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese participants greater than or equal to 20 years of age.
* Diagnosis of chronic, stable plaque psoriasis for at least 6 months prior to screening as defined by: Psoriasis Area Severity Index (PASI) score ≥ 12 and BSA ≥ 10%.
* Psoriasis which is considered inappropriate for topical therapy (based on severity of disease and extent of affected area) or has not been adequately controlled or treated by topical therapy in spite of at least 4 weeks of prior therapy with at least one topical medication for psoriasis or per label.
* In otherwise good health based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry, hematology, immunology, and urinalysis.

Exclusion Criteria:

* Other than psoriasis, history of any clinically significant and uncontrolled systemic diseases; any condition, including the presence of laboratory abnormalities, which would place the participant at unacceptable risk or confound the ability to interpret the data in the study.

Prior medical history of suicide attempt or major psychiatric illness requiring hospitalization within the last 3 years

* Pregnant or breastfeeding.
* History of or ongoing chronic or recurrent infectious disease.
* Active tuberculosis (TB) or a history of incompletely treated TB.
* Clinically significant abnormality on 12-lead ECG or on chest radiograph at screening.
* History of human immunodeficiency virus (HIV) infection or have congenital or acquired immunodeficiencies (eg, Common Variable Immunodeficiency).
* Hepatitis B surface antigen or hepatitis B core antibody positive at screening; positive for antibodies to hepatitis C at screening.
* Malignancy or history of malignancy, except for treated (ie, cured) basal cell or squamous cell in situ skin carcinomas or treated (ie, cured) cervical intraepithelial neoplasia or carcinoma in situ (CIN) of the cervix with no evidence of recurrence within previous 5 years.
* Psoriasis flare within 4 weeks of screening.
* Topical therapy within 2 weeks prior to randomization or systemic therapy for psoriasis or psoriatic arthritis within 4 weeks prior to randomization.
* Use of etretinate within 2 years prior to randomization for females of child bearing potential (FCBP) or within 6 months for males, and within 4 weeks prior to randomization for non-FCBP.
* Use of phototherapy: Ultraviolet light B (UVB), Psoralens and long-wave ultraviolet radiation (PUVA) within 4 weeks prior to randomization or prolonged sun exposure or use of tanning booths or other ultraviolet light sources.
* Use of adalimumab, etanercept, certolizumab pegol, abatacept, tocilizumab, golimumab or infliximab within 12 weeks prior to randomization; use of ustekinumab, alefacept or briakinumab within 24 weeks prior to randomization.
* Any investigational drug within 4 weeks prior to randomization.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (56):
- Japan (56):
  - Ekihigashi Hifuka Clinic, Fukuoka, Fukuoka
  - Tsutsui Clinic Dermatology & Plastic Surgery, Fukuoka, Fukuoka
  - Yano Hifuka Hinyokika Clini, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - HATAMOTO Derma Clinic, Fukuoka, Fukuoka
  - Tomoko Matsuda Dermatological Clinic, Fukuoka, Fukuoka
  - TASHIRO Dermatological Clinic, Iizuka-shi, Fukuoka
  - Okubo Skin Care and Clinic, Itoshima-shi, Fukuoka
  - Matsuda Dermatology Clinic For Skin, Hair, Nail Diseases, Itoshima-shi, Fukuoka
  - Kitakyushu Municipal Medical Center, Kitakyushu, Fukuoka
  - Kyushu Kosei Nenkin Hospital, Kitakyushu, Fukuoka
  - Kyusyu Rosai Hospital, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Matsuo Clinic, Nishiku, Fukuoka
  - Yame General Hospital, Yame, Fukuoka
  - Kokubu Medical Office Abashiri Dermatology Clinic, Abashiri-shi, Hokkaido
  - Chitose Dermatology Plastic Surgery Clinic, Chitose-shi, Hokkaido
  - Asanuma Dermatology Clinic, Chitose-shi, Hokkaido
  - Kokubu Dermatology, Kitami-shi, Hokkaido
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Fukuzumi Dermatology Clinic, Sapporo, Hokkaido
  - Kobe City Medical Center, Kobe, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Teikyo University School of Medicine University Hospital, Kawasaki, Kanagawa
  - Kawasaki Saiwai Clinic, Kawasaki-shi, Kanagawa
  - Sagamihara National Hospital, Sagamihara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Queen's Square Medical Facilities, Yokohama, Kanagawa
  - Nomura Dermatology Clinic, Yokohoma City, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Kosumi lin, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto, Kumamoto
  - Kume Derma Clinic, Sakai-Shi, Osaka
  - SANRUI Dermatology, Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Sugai Dermatologist Park Side Clinic, Utsunomiya, Tochigi
  - Kayaba Dermatology Clinic, Cyu-o-ku, Tokyo
  - Tokai University School of Medicine, Hachiōji, Tokyo
  - Inagi Municipal Hospital, Inagi, Tokyo
  - TSUTSUMI Clinic, Itabasi-Ku, Tokyo
  - Koto Hospital, Koto-ku, Tokyo
  - Maruyama Dermatology Clinic, Koto-ku, Tokyo
  - OIZUMI HANAWA Clinic, Nerima-ku, Tokyo
  - Kitahara Dermatology Clinic, Setagaya-ku, Tokyo
  - NAOKO Dermatology Clinic, Setagaya-ku, Tokyo
  - Mita Dermatology Clinic, Shiba Minato-k, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjyuku-ku, Tokyo
  - Taneda Dermatology Clinic, Suginami-ku, Tokyo
  - Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tachikawa, Tokyo
  - Shakaihoken Simonoseki Kosei Hospital, Shimonoseki-shi, Yamaguchi
  - Matsuo Clinic, Fukuoka
  - AMC Nishiumeda Clinic, Osaka
  - Tokyo Center Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Ohtsuki M, Okubo Y, Komine M, Imafuku S, Day RM, Chen P, Petric R, Maroli A, Nemoto O. Apremilast, an oral phosphodiesterase 4 inhibitor, in the treatment of Japanese patients with moderate to severe plaque psoriasis: Efficacy, safety and tolerability results from a phase 2b randomized controlled trial. J Dermatol. 2017 Aug;44(8):873-884. doi: 10.1111/1346-8138.13829. Epub 2017 Apr 9. PMID 28391657
- [Background] Ohtsuki M, Kubo H, Morishima H, Goto R, Zheng R, Nakagawa H. Guselkumab, an anti-interleukin-23 monoclonal antibody, for the treatment of moderate to severe plaque-type psoriasis in Japanese patients: Efficacy and safety results from a phase 3, randomized, double-blind, placebo-controlled study. J Dermatol. 2018 Sep;45(9):1053-1062. doi: 10.1111/1346-8138.14504. Epub 2018 Jun 15. PMID 29905383
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have had a diagnosis of chronic, stable plaque psoriasis at least 6 months prior to screening and which was considered inappropriate for topical therapy (e.g, based on the severity of the disease and extent of affected area) or could not be adequately controlled/treated with topical therapy to qualify for the study.
Pre-assignment Details: Treatment assignments were stratified according to whether the participants had a psoriatic arthritis (PsA) diagnosis by Classification Criteria for Psoriatic Arthritis (CASPAR) criteria (yes/no) at screening, whether they participated in the sparse pharmacokinetic (PK) sampling, and whether they had participated in the intensive PK sampling.
Groups:
- Placebo: Participants who were initially randomized to identically matching placebo (PBO) by mouth (PO) twice a day (BID) during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20 mg: Participants were randomized to apremilast 20 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) and remained on apremilast 20 mg PO BID dosing during the active treatment phase (weeks 16-68).
- Apremilast 30 mg: Participants were randomized to apremilast 30 mg PO BID during the Placebo-controlled Phase (Weeks 0-16) and remained on apremilast 30 mg PO BID dosing during the active treatment phase (weeks 16-68).
- Placebo-Apremilast 20 mg: Participants who were initially randomized to identically matching PBO PO BID during the Placebo-controlled Phase (weeks 0-16) were re-randomized to apremilast 20 mg PO BID and remained on apremilast 20 mg PO BID dosing during the active treatment phase (weeks 16-68).
- Placebo-Apremilast 30 mg: Participants who were initially randomized to identically matching PBO PO BID during the Placebo-controlled Phase (weeks 0-16) were re-randomized to apremilast 30 mg PO BID and continued dosing with apremilast 30 mg PO BID during the active treatment phase (weeks 16-68).
Period: Placebo-Controlled Phase Week 0-16
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo-Apremilast 20 mg | Placebo-Apremilast 30 mg
Started | 84 | 85 | 85 | 0 | 0
Completed | 72 | 69 | 76 | 0 | 0
Not Completed | 12 | 16 | 9 | 0 | 0
Not completed — Adverse Event | 3 | 10 | 6 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 1 | 0 | 0
Period: Active Treatment Phase (Weeks 16-68)
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo-Apremilast 20 mg | Placebo-Apremilast 30 mg
Started | 0 | 69 | 76 | 36 | 35
Completed | 0 | 56 | 65 | 33 | 30
Not Completed | 0 | 13 | 11 | 3 | 5
Not completed — Adverse Event | 0 | 6 | 3 | 3 | 2
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 4 | 0 | 1
Not completed — Principal Investigator Signature Missing | 0 | 1 | 2 | 0 | 2
Period: Observational Follow-up Phase
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Placebo-Apremilast 20 mg | Placebo-Apremilast 30 mg
Started | 12 | 82 | 83 | 36 | 33
Completed | 12 | 79 | 82 | 36 | 33
Not Completed | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat Population = (mITT) population consisted of all participants who were randomized and received at least one dose of investigational product (IP). Participants were included in the treatment group in which they were randomized.
Groups:
- Placebo: Participants initially randomized to identically matching placebo during the 16-week placebo controlled phase.
- Apremilast 20 mg: Participants initially randomized to apremilast 20mg BID during the 16-week placebo controlled phase.
- Apremilast 30 mg: Participants initially randomized to apremilast 30mg BID during the 16-week placebo controlled phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg | Total
Number analyzed (Participants) | 84 | 85 | 85 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.98) | 52.2 (12.54) | 51.7 (12.73) | 50.8 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 14 | 52
  Male | 62 | 69 | 71 | 202
Region of Enrollment [Number; unit: Participants]
  Japan | 84 | 85 | 85 | 254

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a 75% Improvement (Response) From Baseline in the Psoriasis Area and Severity Index (PASI-75) at Week 16
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement was missing.
Time Frame: Baseline to Week 16
Population: mITT consisted of all participants who were randomized and received at least one dose of IP. Participants were included in the treatment group in which they were randomized. Missing values were imputed using the Last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 20mg: Participants initially randomized to apremilast 20mg BID during the 16-week placebo controlled phase.
- Apremilast 30mg: Participants initially randomized to apremilast 30mg BID during the 16-week placebo controlled phase.
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
percentage of participants | 7.1 | 23.5 | 28.2
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0032, Chi-squared; Difference = 16.4, 95% CI 2-sided [5.8 to 27.0]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p = 0.0003, Chi-squared; Difference = 21.1, 95% CI 2-sided [10.1 to 32.1]

2. Secondary Outcome: Percentage of Participants Who Achieved a Static Physician's Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) With at Least 2 Point Reduction From Baseline to Week 16
Description: The sPGA is a measure of psoriasis disease severity at the time of evaluation by the Investigator. It does not compare assessments across visits or rely on investigator recall or prior disease. The sPGA is a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (severe; majority of plaques have severe thickness, erythema, and scaling). The investigator examines all of the lesions on the participant and assigns a score ranging from 0 to 5 for thickness, erythema and degree of scaling. Scores for thickness, erythema and scaling are then summed and the mean of these 3 scores equals the overall sPGA score.
Time Frame: Baseline to Week 16
Population: mITT population with a sPGA greater than 2 at baseline. Participants were included in the treatment group in which they were randomized. Missing values were imputed using the LOCF method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 68 | 71 | 71
percentage of participants | 8.8 | 23.9 | 29.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0165, Chi-squared; Difference = 15.1, 95% CI 2-sided [3.1 to 27.1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p = 0.0020, Chi-squared; Difference = 20.8, 95% CI 2-sided [8.2 to 33.3] — Missing values were imputed using the LOCF method

3. Secondary Outcome: Percent Change From Baseline in the Psoriasis Affected Body Surface Area (BSA) at Week 16
Description: BSA is a measurement of involved skin. The overall BSA affected by psoriasis is estimated based on the palm area of the subject's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area.
Time Frame: Baseline to Week 16
Population: mITT population consisted of all participants who were randomized and received at least one dose of IP. Participants were included in the treatment group in which they were randomized. Missing values were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
percent change | 7.5 (5.56) | -21.6 (5.52) | -30.5 (5.51)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -29.1, 95% CI 2-sided [-44.5 to -13.6] — 2-sided 95% CI and p-values were based on an analysis of covariance model with treatment arm as a factor and baseline value as a covariate. Means (LS Means) and p-values were adjusted by covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -38.0, 95% CI 2-sided [-53.4 to -22.6] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in the Psoriasis Area and Severity Index (PASI) Score
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. The PASI is a validated instrument that has become standard in clinical trials for psoriasis. The PASI scores range from 0 to 72, with higher scores reflecting a greater disease severity.
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
percent change | -3.7 (5.55) | -33.1 (5.51) | -43.1 (5.50)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -29.5, 95% CI 2-sided [-44.9 to -14.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -39.5, 95% CI 2-sided [-54.9 to -24.1] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants Who Achieved a 50% Improvement From Baseline (Response) Reduction in the PASI-50 at Week 16
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement is missing.
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
percentage of participants | 21.4 | 41.2 | 50.6
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0057, Chi-squared; Difference = 19.7, 95% CI 2-sided [6.1 to 33.4]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 29.2, 95% CI 2-sided [15.4 to 42.9]

6. Secondary Outcome: Change From Baseline in Pruritus Visual Analogue Scale 100-mm (VAS) at Week 16
Description: The pruritus visual analog scale (VAS) was used to measure the amount of itching and discomfort a participant experiences. Participant's assessment of pruritus (Itch) asked: On average, how much itch have you had because of your condition in the past week? Higher scores correspond to more severe symptom or disease. The participant places a vertical line on a 100-mm VAS on which the left-hand boundary represents no itch at all and the right-hand boundary represents the worst itch imaginable. The distance from the vertical line to the left-hand boundary is recorded. VAS scores range from 0 to 100 mm, where higher scores correspond to worse pruritis (itch).
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
units on a scale | 7.1 (2.86) | -7.5 (2.84) | -17.7 (2.83)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -14.6, 95% CI 2-sided [-22.6 to -6.7] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -24.8, 95% CI 2-sided [-32.7 to -16.9] — 2-sided 95% CI and p-values were based on an analysis of covariance model with treatment arm as a factor and baseline value as a covariate. Means (LS Means) and p-values were adjusted by covariate. Missing values were imputed using the LOCF method

7. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16
Description: Dermatology Life Quality Index (DLQI) was developed as a practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains 10 items dealing with the participants skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score has a possible range from 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
units on a scale | 1.3 (0.53) | -0.5 (0.53) | -2.2 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.0204, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.2 to -0.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-4.9 to -2.0] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Change From Baseline in Mental Component Summary (MCS) Score of the Medical Outcome Study Short Form 36-item (SF-36) Health Survey Version 2.0 at Week 16
Description: SF-36 is a 36-item general health status instrument often used in clinical trials and health services research. It consists of 8 scales: physical function (PF), role limitations-physical (RP), vitality (VT), general health perceptions (GH), bodily pain (BP), social function (SF), role limitations-emotional (RE), and mental health (MH). Scale scores range from 0 to 100, with higher scores indicating better quality of life (better functioning)
Time Frame: Baseline to Week 16
Population: mITT population consisted of all participants who were randomized and received at least one dose of IP. Participants were included in the treatment group in which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
units on a scale | -1.59 (0.953) | -0.71 (0.953) | 0.27 (0.948)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 20mg; Test type: Superiority or Other; p = 0.5149, ANCOVA; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-1.78 to 3.53] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 30mg; Test type: Superiority or Other; p = 0.1693, ANCOVA; Mean Difference (Final Values) = 1.85, 95% CI 2-sided [-0.79 to 4.50] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Number of Participants Who Achieved an American College of Rheumatology Criteria (ACR) 20% Improvement (ACR 20)
Description: The ACR 20 is defined as a 20% improvement in joint tenderness (78 joint count) and joint swelling scores (76 joint count) compared to baseline plus 20% improvements in 3 of the following 5 assessments (compared to baseline): subject global assessment of disease activity (measured on a 100-mm visual analog scale [VAS]); physician global assessment of disease activity (measured on a 100-mm VAS); subject self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI] score); subject assessment of pain (measured on a 100-mm VAS); and CRP level.
Time Frame: Baseline to Week 16
Population: Due to the small sample size in the study for the ACR 20 % improvement, the analysis was not conducted. The decision not to perform the analysis was authorized by the lead therapeutic executive and there is no data available to analyze. No resources are available to conduct the ACR 20% improvement endpoint for this population.
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Percent Change From Baseline Psoriatic Arthritis Pain Visual Analogue Scale (VAS)
Description: Change from baseline in psoriatic arthritis pain 100-mm VAS; The participant places a vertical line on a 100-mm VAS on which the left-hand boundary represents no pain at all and the right-hand boundary represents the worst possible pain. The distance from the vertical line to the left-hand boundary is recorded.
Time Frame: Baseline to Week 16
Population: Due to the small sample size in the study for change from baseline in psoriatic arthritis pain VAS, the analysis was not conducted. The decision not to perform the analysis was authorized by the lead therapeutic executive and there is no data to analyze. No resources are available to conduct the analysis for the end point.
Groups:
- Apremilast 20 mg: Participants initially randomized to apremilast 20mg PO BID during the 16-week placebo controlled phase.
- Apremilast 30 mg: Participants initially randomized to apremilast 30mg PO BID during the 16-week placebo controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Percent Change From Baseline in Physical Function Assessment Using the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Change from baseline in physical function assessment using HAQ-DI; The HAQ-DI is a 20-question, self-administered instrument that measures the subject's functional ability on a 4-level difficulty scale (0-3, with 0 representing normal or no difficulty; and 3 representing inability to perform). Eight categories of functioning are included: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities.
Time Frame: Baseline to Week 16
Population: Due to the small sample size for the change from baseline in physical function assessment using the HAQ-DI, the analysis was not conducted. The decision not to perform the analysis was authorized by the lead therapeutic executive and there is no data available to analyze. No resources are available to conduct the analysis for the end point.
Groups:
- Placebo: Participants initially randomized to identically matching placebo PO BID during the 16-week placebo controlled phase.
Arm/Group | Placebo | Apremilast 20 mg | Apremilast 30 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AE) in the Placebo Controlled Phase
Description: An AE was any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: Baseline to Week 16
Population: Safety population consisted of all participants who were randomized and received at least one dose of IP
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 84 | 85 | 85
participants
  ≥ At least 1 TEAE | 35 | 49 | 44
  ≥ 1 Drug-related TEAE | 8 | 18 | 25
  ≥ At least 1 Severe TEAE | 1 | 4 | 0
  ≥ 1 Serious TEAE | 0 | 4 | 0
  Any Serious Drug-related TEAE | 0 | 2 | 0
  ≥ 1 TEAE leading to Drug Interruption | 2 | 2 | 0
  ≥ 1 TEAE Leading to Drug Withdrawal | 4 | 10 | 6
  ≥ 1 TEAE Leading to Death | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events (AE) in the During the Apremilast-exposure Period
Description: An AE was any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above. An AE is a treatment emergent AE if the AE start date is on or after the date of the first dose of study drug and no later than 28 days after the last dose.
Time Frame: From the first dose of apremilast (either Week 0 or Week 16 for participants originally randomized to placebo who were re-randomized at Week 16) until 28 days after the last dose of apremilast.
Population: All participants who received apremilast at any time during the trial.
Measure: Number; unit: participants
Groups:
- Apremilast 20mg: Participants who received their first dose of apremilast 20 mg PO BID during the placebo-controlled phase or those who were originally randomized to placebo and were subsequently re-randomized to apremilast 20 mg PO BID.
- Apremilast 30mg: Participants who received their first dose of apremilast 30 mg PO BID during the placebo-controlled phase or those who were originally randomized to placebo and were subsequently re-randomized to apremilast 30 mg PO BID.
Arm/Group | Apremilast 20mg | Apremilast 30mg
Number analyzed (Participants) | 121 | 120
participants
  ≥ At Least 1 TEAE | 94 | 89
  ≥ 1 Drug-related TEAR | 34 | 37
  ≥ At Least 1 Severe TEAE | 12 | 2
  ≥ 1 Serious TEAE | 11 | 2
  Any Serious Drug-related TEAE | 5 | 0
  ≥ 1 TEAE leading to Drug Interruption | 6 | 2
  ≥ 1 TEAE Leading to Drug Withdrawal | 19 | 10
  ≥ 1 TEAE Leading to Death | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs are reported for the 16-week placebo-controlled phase and up to 68 weeks for those who received apremilast during the study; TEAEs were recorded from the date of the first dose of IP received to no later than 28 days after the last dose of IP
Groups:
- Placebo (Weeks 0-16): Participants initially randomized to identically matching placebo (PBO) by mouth (PO) twice a day (BID) during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20mg BID (Weeks 0-16): Participants initially randomized to receive apremilast 20 mg BID PO during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 30mg BID (Weeks 0-16): Participants initially randomized to apremilast 30 mg BID PO during the Placebo-controlled Phase (Weeks 0-16).
- Apremilast 20mg BID (Weeks 0-68): Participants who received 20 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 16 up until Week 68.
- Apremilast 30mg BID (Weeks 0-68): Participants who received 30 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 16 up until Week 68
Arm/Group | Placebo (Weeks 0-16) | Apremilast 20mg BID (Weeks 0-16) | Apremilast 30mg BID (Weeks 0-16) | Apremilast 20mg BID (Weeks 0-68) | Apremilast 30mg BID (Weeks 0-68)
Serious Adverse Events (participants affected / at risk) | 0/84 | 4/85 | 0/85 | 11/121 | 2/120
Other Adverse Events (participants affected / at risk) | 9/84 | 16/85 | 18/85 | 35/121 | 40/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=84) | Apremilast 20mg BID (Weeks 0-16) (N=85) | Apremilast 30mg BID (Weeks 0-16) (N=85) | Apremilast 20mg BID (Weeks 0-68) (N=121) | Apremilast 30mg BID (Weeks 0-68) (N=120)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-16) (N=84) | Apremilast 20mg BID (Weeks 0-16) (N=85) | Apremilast 30mg BID (Weeks 0-16) (N=85) | Apremilast 20mg BID (Weeks 0-68) (N=121) | Apremilast 30mg BID (Weeks 0-68) (N=120)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 6 | 3 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 8 | 10 | 12
Nasopharyngitis (Infections and infestations) | 7 | 10 | 10 | 28 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 12 months since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.